CLINICAL TRIAL: NCT06542653
Title: Effect of PCI on Clinical Prognosis of Chronic Coronary Artery Occlusion
Status: Recruiting | Type: Observational
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Chen Leilei, Director, The First Affiliated Hospital with Nanjing Medical University
Other Study IDs: CTO-PCI
Record Dates: First submitted 2024-08-01; First posted 2024-08-07 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Coronary Atheroscleroses
Keywords: Chronic total occlusion; Percutaneous coronary intervention; Major adverse cardiovascular events
MeSH Terms: conditions — Coronary Artery Disease | interventions — Percutaneous Coronary Intervention

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- CTO-PCI group: successful percutaneous coronary intervention (PCI)
  Interventions: Procedure: PCI; Drug: OMT
- CTO-OMT group: optimal medical therapy (OMT)
  Interventions: Drug: OMT

INTERVENTIONS:
Procedure: PCI — successful percutaneous coronary intervention (PCI) in Coronary chronic total occlusions (CTOs) patients
  Other Names: percutaneous coronary intervention
  Groups: CTO-PCI group
Drug: OMT — optimal medical therapy (OMT) in CTO patients, such as aspirin 1td, ACEI/ARB 1td, β blocker 1td, statin 1td.
  Other Names: optimal medical therapy

SUMMARY:
Coronary chronic total occlusions (CTOs) are considered to increase the risk of adverse clinical outcomes. The purpose of this study was to evaluate whether long-term clinical outcomes could be improved by successful percutaneous coronary intervention (PCI) over optimal medical therapy (OMT) in CTO patients.

DETAILED DESCRIPTION:
patients with CTO lesions undergoing PCI at the First Affiliated Hospital of Nanjing Medical University from January 2011 to December 2017 were enrolled. After someone were excluded due to CABG surgery, patients who met the enrollment criteria were divided into successful CTO-PCI group and CTO-OMT group based on the treatment received. The study primary endpoint was major adverse cardiac cerebrovascular events (MACCE), including cardiac death, recurrent myocardial infarction, unplanned revascularization, and stroke. The secondary endpoint was all-cause death.

ELIGIBILITY:
Inclusion Criteria:

* patients with at least one coronary CTO lesion at our hospital in between January 2011 and December 2017

Exclusion Criteria:

* (1) patients with ST-segment elevation myocardial infarction (STEMI)
* (2)a history of coronary artery bypass grafting (CABG)
* (3) cardiogenic shock
* (4) malignant tumor. Patients were referred for PCI based on CTO-related symptoms or evidence of viability, or corresponding ischemia in the area of the CTO artery.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients were referred for PCI based on CTO-related symptoms or evidence of viability, or corresponding ischemia in the area of the CTO artery. The enrolled patients were divided into 2 groups, i.e., CTO-PCI group (n=187) and CTO-OMT group (n=46). The strategy to perform PCI on CTO patients was dependent on some factors, including co-morbidity, technical challenges, operators' preference
Sampling Method: Non-Probability Sample
Enrollment: 258 (Estimated)
Dates: Start 2023-09-17 (Actual); Primary Completion 2024-09-17 (Actual); Study Completion 2025-09-17 (Estimated)

PRIMARY OUTCOMES:
major adverse cardiac cerebrovascular events (MACCE) | January 2011 to December 2023
  including cardiac death, recurrent myocardial infarction, unplanned revascularization, and stroke.

SECONDARY OUTCOMES:
all-cause death | January 2011 to December 2023
  all-cause death

CONTACTS AND LOCATIONS:
Overall Officials: Leilei Chen, Study Director — The First Affiliated Hospital with Nanjing Medical University
Locations (1):
- The First Affiliated Hospital with Nanjing Medical University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided